CLINICAL TRIAL: NCT06415500
Title: A Single Center, Open, Single Arm Clinical Study on the Safety and Preliminary Efficacy of NK042 in the Treatment of Malignant Ascites
Brief Title: A Study on the Safety and Preliminary Efficacy of NK042 in the Treatment of Malignant Ascites
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK042-IIT-MA
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Cancer
Keywords: malignant ascites
MeSH Terms: interventions — NK Cell Lectin-Like Receptor Subfamily B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK042 (Experimental)
  Interventions: Drug: NK042

INTERVENTIONS:
Drug: NK042 — NK042 intraperitoneal infusion on Days 0,7 and 14.
  Other Names: NKR-NK

SUMMARY:
The purpose of this study is to assess the safety and efficacy of NK042 for treatment of malignant ascites.

DETAILED DESCRIPTION:
This is a phase 1 ,open-label , Single Arm,dose escalation study to evaluate the safety, tolerability, PK, PD and preliminary efficacy of NK042 in patients with treatment of malignant ascites caused by Gynecologic Cancer.About 3-9 subjects are planned to be enrolled, Subjects will receive intraperitoneal infusion of NK042 once a week (D0、D7、D14)for 2 cycles, with 3 times during each cycle and a total of 6 infusions. The occurrence of DLTs will be observed from the first intraperitoneal infusion of NK042 to 28 days after infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have the ability to know and sign informed consent;
2. Age 18-70 years old; any sex;
3. Histologically or pathologically confirmed Gynecologic Cancer,including but are not limited to patients with malignant ascites caused by advanced malignant tumors such as ovarian cancer and endometrial cancer;
4. The volume of ascites ≥1L based on CT or more than the same amount of abdominal fluid (definition: abdominal fluid ≥4.5cm detected by B ultrasound in lying position, accompanied by clinical symptoms such as abdominal distension and discomfort);
5. Ascites should be treated by puncture;
6. Expected survival time ≥ 12 weeks;
7. the Eastern Cooperative Oncology Group (ECOG) scored 0-2 points;
8. Appropriate organ and bone marrow function,Laboratory test results must meet the following criteria(unless otherwise specified, the test results of the research center shall prevail)： (1)blood routine examination: White blood cell count > 3×10^9/L; Absolute neutrophil Count (ANC)≥1.5×10^9/L; Haemoglobin > 90 g/L; lymphocyte count ≥ 0.7×10^9/L; Platelet count ≥ 75×10^9/L. (2)renal function: Serum creatinine and/or urea < 1.5×ULN; serum total bilirubin (TBIL) ≤ 1.5 × Upper limit of normal value (ULN)(bilirubin ≤ 3×ULN for patients with Gilbert's syndrome; (3)liver function: ALT and AST ≤ 2.5 × ULN(≤ 5×ULN for patients with complication of liver metastases);
9. Fertility capable subjects (male and female) must agree to use reliable;contraceptive methods (hormone or barrier methods or abstinence) during the trial and at least 1 year after the last dose; Female subjects of reproductive age must have a negative blood or urine pregnancy test within 14 days before enrollment;
10. For previous anti-malignant ascites therapy (except systemic chemotherapy to control the primary tumor), the washout period is set to 2 weeks or 5 half-lives after the end of the last dose, whichever is shorter;
11. The subjects were able to communicate well with the researchers, and understand and comply with the requirements of this trial.

Exclusion Criteria:

1. Currently, or within 30 days prior to enrollment, participating in a clinical trial of another drug or biologic therapy, or having received comparable cellular therapy;
2. Patients undergoing treatment for intraperitoneal malignant ascites, including therapeutic paracentesis;
3. Systemic or other treatments that have a significant impact on the evaluation of efficacy are determined according to the study;
4. Patients with extensive liver metastases Patients with extensive liver metastases (tumor volume occupying approximately >70% of total liver volume);
5. Occurrence of complete intestinal obstruction within 30 days before the first dose, or diagnosis of incomplete intestinal obstruction deemed unsuitable for participation in the trial based on symptoms and signs as determined by the investigator;
6. Laboratory results indicating bacterial peritonitis (neutrophil count > 250 / µl ascites);
7. Serum albumin ≤ 30 g/L;
8. Meet any of the following criteria related to cardiac function: 1) Various clinical significant arrhythmia or conduction abnormalities that require clinical intervention; 2) Congenital QT interval prolongation syndrome or men with QTc>450 msec and women with QTc>470 msec (QTc is calculated using Fridericia's correction formula), or taking drugs that may cause QT interval prolongation or torsade de pointe arrhythmia; 3) Various clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina pectoris, coronary artery bypass surgery or peripheral artery bypass grafting surgery, and cerebrovascular events (referring to thromboembolic or hemorrhagic cerebrovascular events, excluding cerebrovascular events caused by anemia caused by underlying disease ) within the first 6 months of enrollment, congestive heart failure with a New York Heart Association (NYHA, Attachment 8) rating of 3 or higher, or a left ventricular ejection fraction (LVEF) of<50%;
9. Subjects with chronic or relapsed severe autoimmune or immune-mediated disease requiring high-dose steroid or other immunosuppressive therapy;
10. The presence of central nervous system (CNS) metastases is known;
11. Subjects with active systemic infections requiring treatment, including, but not limited to, subjects with active tuberculosis, subjects with Hepatitis B Surface Antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb) positivity and peripheral blood HBV DNA titers greater than the upper limit of detection, subjects who are RNA positive for Hepatitis C (HCV), subjects who are seropositive for Human Immunodeficiency Virus (HIV), subjects who are seropositive for Helicobacter syphilis, etc.; and Subjects who are seropositive for Hepatitis C (HCV);
12. Subjects who have previously undergone liver transplantation, organ allograft transplantation, or renal replacement therapy;
13. Active lung disease, including but not limited to interstitial lung disease or pneumonia (except for local interstitial pneumonia induced by radiotherapy), pulmonary fibrosis, etc;
14. Meet any of the following criteria, 1) history of abuse of psychotropic substances and unable to abstain or with mental disorders, 2) have a serious concomitant disease that endangers the safety of the patient or affects the completion of the trial judged by the researcher;
15. Women during pregnancy or lactation;
16. Hypersensitivity to albumin, DMSO;
17. Co-existing HBV and HCV and two or more viral infections;
18. The researcher judge the patient with factors that may affect the results of the study or interfere the participation in the entire study process, including but not limited to previous or existing physical conditions, treatment or laboratory abnormalities, etc; Or putting the patient in a high-risk situation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose-limiting Toxicity (DLT) | 28 Days
  The occurrence of DLTs will be observed from the first intraperitoneal infusion of NK042 to 28 days after infusion.

SECONDARY OUTCOMES:
ascites volume | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  Five-point method to measure ascites volume(base on CT).
Time to next therapeutic puncture，TTpu | From the time of first dosing (Day 1) to the next puncture/drainage (up to 6 months)
  The time to the next puncture/drainage
Puncture-free survival, PuFS | From the time of of first dosing (Day 1) to the next puncture/drainage or death (up to 6 months)
  The time to the next puncture/drainage or death
Progression-free Survival, PFS | From the time of first dosing (Day 1) until disease progression or toxicity intolerance or death (up to 6 months).
  The time to disease progression assessed by the imaging evaluation or toxicity or death
Overall survival, OS | From the time of first dosing (Day 1) until death (up to 6 months).
  The time to death

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No